## Mr D Lawrie **Consultant Orthopaedic Surgeon Upper Limb Unit Department of Orthopaedics** Woodend Hospital, Eday Road, Woodend, Aberdeen, AB15 6XS



**Study Title:** Comparison Two Treatment of Dorsal Wrist Ganglia;

Aspiration alone vs Aspiration and Injection of Platelet Rich Plasma

**Participant ID Number:** 

**Chief Investigator:** David Lawrie **IRAS ID:** 205497

Version: 5 - 03/06/2018

## **CONSENT FORM**

| | | Please | initiai bo |
|---|---|---|---|
| 1 | I confirm that I have read and understand the information sheet Version No: < <i>Current version No&gt;</i> Date: < <i>Current version date&gt;</i> for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily | | |
| 2 | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | | |
| 3 | I understand that relevant sections of my medical notes and data collected during study may be looked at by individuals from NHS Grampian or from regulatory authorities if appropriate, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | |
| 4 | I agree to my GP being informed of my participation in the study. | | |
| 5 | I understand de-identified data will be collected, stored and analysed by Arthrex using Surgical Outcomes System. | | |
| 6 | I agree for my information to be stored on NHS Grampian servers. | | |
| 7 | I agree to take part in the above study. | | |
| 8 | I agree to under go injection with platelet rich plasma injection if I am selected for that arm of the study. | | |
| Name of Patient Date Signature | | Signature | |
| | Name of Person taking consent Date if different from researcher) | Signature | |
| Re | Researcher Date | Signature | <del></del> |

1 for patient; 1 for researcher; 1 to be kept with hospital notes